CLINICAL TRIAL: NCT01847729
Title: A Multicenter Study Assessing the Prevalence of Co-addictions in Subjects Receiving Maintenance Treatment for Opiate Dependence. Determination of Clinical and Pharmacological Profil.
Brief Title: OPAL: "Opiates and PhArmacoLogy"
Acronym: OPAL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0498
Record Dates: First submitted 2013-04-10; First posted 2013-05-07 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Substance Use Disorder
Keywords: Opiate dependence; Opiate substitution treatment; co-addictions; Patients addicted to opiates; methadone; buprenorhine; morphine; OST in place; pathological gambling; pharmacokinetic; pharmacogenetic; polymorphism; cytochrome P450 2D6; Therapeutic Drug Monitoring
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Gambling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting 2 EDTA tubes of 5 mL (blood)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients on OST prescribed to treat opiate dependence: Collecting socio-demographic data, data concerning opiate dependence, data about other substance use disorder, data regarding gambling practice, psychopathological data.

SUMMARY:
The aim of this study is to determine the current prevalence of co-addictions, including problem/pathological gambling, in patients receiving Opiate Substitution Treatment (OST), and to then compare patients receiving OST with or without a co-addiction (excluding tobacco dependence) in order to determine their clinical profile.

In addition, an ancillary study to be carried out only among those patients receiving methadone, will aim to etablish whether a low plasma concentration of methadone, on the one hand, and an ultrarapid metabolizer genetic profile, on the other, are the characteristics most commonly associated with the presence of co-addictions. This will allow us to complete patient's pharmacological characterization.

DETAILED DESCRIPTION:
Non-interventionel study Total duration: 12 months (preparation, recruitment, analysis) Recruitment period: 6 months Duration of monitoring per patient: no monitoring

Main objective: to assess the current prevalence of addictive co-morbidities in opiate-dependent subjects receiving Opiate Substitution Treatment (OST) for at least 6 months.

Secondary objective: to compare patients being treated using OST who currently have a co-addiction (with the exception of tobacco dependence) with patients being treated with OST who do not currently have a co-addiction, based on pharmacological and clinical characteristics (for pharmacological characteristics: pharmacokinetic and pharmacogenetic analyses as part of an ancillary study into only those patients being treated with methadone).

Main judgment criterion: Presence or absence of co-addictions (except tobacco dependence), determined using assessment tools.

The secondary assessment criteria shall be: sociodemographic data, data about opiate dependence, data about other substance use disorders, data about gambling practice, psychopathological data (impulsivity, ADHD), pharmacokinetic data and pharmacogenetic data.

Statistical analysis: For the main judgment criterion, a rate of prevalence of current co-addictions will be estimated using a 95% confidence interval.

Descriptive analyses will be carried out for all variables gathered and along with point estimates and 95% confidence intervals for qualitative and quantitative variables.

The second stage will involve univariate exploratory analyses. The two groups of patients will be compared according to the presence or absence of co-addictions. For the quantitative variables Student tests or non parametric tests will be used. For the qualitative variables, we will use Chi-squared or Fisher tests.

Finally, multivariate analyses will be carried out. The factors that have been previously identified as a being linked to co-addictions (with the threshold p = 0.2) will the be incorporated into logistic regression models. The best model, wich enables explanation of the co-addictions will then be selected using likelihood ratio tests.

ELIGIBILITY:
General Inclusion Criteria:

* Over 18,
* Under treatment unsing methadone or buprenorhine (+/- naloxone) or morphine as substitute, prescribed for opiate dependence,
* OST begining at least 6 months previously,
* Incarceration for less than a month in the event of monitoring in SMPR,
* Good understanding of French, able to read and write.

General non-Inclusion Criteria:

* Protected adults (guardianship, wardship)
* Disorder of higher-order brains functions (severe cognitive disorders or confusion) or psychotic disorder (hallucinations, delusion) that may interfere with the study.

Non-Inclusion criteria for patients participating in the ancillary study:

* Medical monitoring by a doctor from the Drug Addiction Network of the Nantes Area,
* OST other than methadone
* Adjustement to dosage in the 5 days prior to administering OST
* Pregnant women
* Absence of social security registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study deals with patients on OST precsribed to treat opiate dependence; the OST may be methadone, buprenorphine (+/- naloxone) or a morphine-based drug.
  The total group of patients to be inclued is estimated at 384 patients. Of these patients, 200 will take part in the ancillary study.
  The number of recruitment centers foreseen allows this objective to be met in 6 months.
  Those participating in this study will not be able to participate in another study (notably in order to avoid drug interactions).
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Presence or absence of co-addictions (exept tobacco dependence) | 1 day
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marie Grall-Bronnec, PH, Study Director — Nantes University Hospital; Régis Bouquié, AHU, Principal Investigator — Nantes University Hospital; Stéphane Bézieau, Pr, Principal Investigator — Nantes University Hospital; Pierre Bodenez, Principal Investigator — University Hospital, Brest; Morgane Guillou-Landréat, Principal Investigator — Morlaix Hospital; Bertrand Legeay, Principal Investigator — Medico-psychological regional service nantes University Hospital; Isabelle Martineau, Principal Investigator — La Métairie center care support and prevention of addiction; Philippe Levassor, Principal Investigator — La Rose des Vents center care support and prevention of addiction; Jean-Yves Guillet, Principal Investigator — General practitioners in the drug-addiction network of the Nantes Area
Locations (7):
- France (7):
  - Brest Universit Hospital, Brest
  - CSAPA "La métairie", La Roche-sur-Yon
  - Morlaix Hospital, Morlaix
  - CSAPA "Le triangle", Nantes
  - University Hospital Nantes, Nantes
  - CSAPA-CAARUD "La rose des vents", Saint-Nazaire
  - Réseau toxicomanie de la région nantaise, Saint-Sébastien-sur-Loire

REFERENCES:
- [Background] Bouju G, Hardouin JB, Boutin C, Gorwood P, Le Bourvellec JD, Feuillet F, Venisse JL, Grall-Bronnec M. A shorter and multidimensional version of the Gambling Attitudes and Beliefs Survey (GABS-23). J Gambl Stud. 2014 Jun;30(2):349-67. doi: 10.1007/s10899-012-9356-3. PMID 23334576
- [Background] Grall-Bronnec M, Wainstein L, Feuillet F, Bouju G, Rocher B, Venisse JL, Sebille-Rivain V. Clinical profiles as a function of level and type of impulsivity in a sample group of at-risk and pathological gamblers seeking treatment. J Gambl Stud. 2012 Jun;28(2):239-52. doi: 10.1007/s10899-011-9258-9. PMID 21698341
- [Background] Grall-Bronnec M, Wainstein L, Augy J, Bouju G, Feuillet F, Venisse JL, Sebille-Rivain V. Attention deficit hyperactivity disorder among pathological and at-risk gamblers seeking treatment: a hidden disorder. Eur Addict Res. 2011;17(5):231-40. doi: 10.1159/000328628. Epub 2011 Jun 7. PMID 21654176
- [Derived] Beslot A, Grall-Bronnec M, Balem M, Schreck B, Laforgue EJ, Victorri-Vigneau C, Guillou-Landreat M, Leboucher J; OPAL-Group; Challet-Bouju G, Cabelguen C. ADHD: prevalence and effect on opioid use disorder treatment outcome in a French sample of patients receiving medication for opioid use disorder-the influence of impulsivity as a mediating factor. Harm Reduct J. 2024 Sep 9;21(1):165. doi: 10.1186/s12954-024-01079-7. PMID 39252018
- [Derived] Guillou Landreat M, Dany A, Challet Bouju G, Laforgue EJ, Cholet J, Leboucher J, Hardouin JB; OPAL Group; Victorri Vigneau C, Grall Bronnec M. How do people who use drugs receiving Opioid Medication Therapy perceive their treatment ? A multicentre study. Harm Reduct J. 2022 Mar 28;19(1):31. doi: 10.1186/s12954-022-00608-6. PMID 35346219
- [Derived] Guillou-Landreat M, Dany A, Challet-Bouju G, Laforgue E, Leboucher J, Benoit Hardouin J, Victorri-Vigneau C, Grall-Bronnec M. What Differs between Patients under Methadone and under Buprenorphine for Opioid Use Disorder (OUD) in Daily Clinical Practice in France? A Short Report. Int J Environ Res Public Health. 2021 Feb 3;18(4):1425. doi: 10.3390/ijerph18041425. PMID 33546494